CLINICAL TRIAL: NCT01219803
Title: Dosage-efficacy Relationship Clinical Trial of Ge Gen Qin Lian Decoction
Brief Title: Trial of Different Dosages' Ge Gen Qin Lian Decoction in the Treatment of Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Tong Xiaolin, Professor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20100727
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2; Dose-Response Relationship, Drug
Keywords: Dose-Response Relationship, type 2 diabetes,TCM
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High dose GGQL Decoction (Experimental)
  Interventions: Drug: High Dose GGQL Decoction
- Mild dose GGQL Decoction (Experimental)
  Interventions: Drug: Mild dose GGQL Decoction
- Low dose GGQL Decoction (Experimental)
  Interventions: Drug: Low dose GGQL Decoction
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: High Dose GGQL Decoction — The drug was a kind of decoction extracted by Chinese herbs such as Huanglian etc,5 times thick of low dose GGQL Decoction, 150ml/bag, twice in a day
  Other Names: High Dose Ge Gen Qin Lian Decoction
  Arms: High dose GGQL Decoction
Drug: Mild dose GGQL Decoction — The drug was a kind of decoction extracted by Chinese herbs such as Huanglian etc,3 times thick of low dose GGQL Decoction, 150ml/bag, twice in a day
  Other Names: Mild dose Ge Gen Qin Lian Decoction
  Arms: Mild dose GGQL Decoction
Drug: Low dose GGQL Decoction — The drug was a kind of decoction extracted by Chinese herbs such as Huanglian etc, 150ml/bag, twice in a day
  Other Names: Low dose Ge Gen Qin Lian Decoction
  Arms: Low dose GGQL Decoction
Drug: Placebo — The placebo was a kind of decoction,which including 4.5% low dose GGQL Decoction to feel bitter taste as other drugs, 150ml/bag, twice in a day
  Other Names: placebo of Ge-Gen-Qin-Lian Decoction
  Arms: Placebo

SUMMARY:
Ge Gen Qin Lian Decoction are one kind of Chinese prescription, and previous study showed they had antidiabetic effects on the clinical patients and no obvious toxicity was found. The purpose of this study was to evaluate the efficacy and safety of different dosage of Ge Gen Qin Lian Decoction in the treatment of type 2 diabetic patients and explore relationship of the dosage and effect and the safety of 3 dosages of Ge Gen Qin Lian Decoction.

DETAILED DESCRIPTION:
two hundred and forty primary diabetic patients will be expected to be recruited, which were divided into different groups in a randomized, doubled blind, dose-paralleled-control multi-centre clinical design. The patients were randomly taken with high-dosage(5 times of low-dosage),mild-dosage(3 times of low-dosage), low-dosage,placebo(4.5% of low dosage) by 2 times every day for 12 weeks. Hemoglobin A1c (HbA1c), Fasting plasma glucose (FPG),postprandial 2 hours plasma glucose(2hPG),insulin(0h,1h,2h),syndrome,symptoms,body mass index (BMI),waist circumference (WC) of these groups were measured and analyzed. Some safety indexes such blood and urine and stool routine examination, electrocardiogram (ECG)and liver and kidney function tests were measured and analyzed during the experiment. The treatment period is 12 week.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes mellitus
* 30-65 years old
* HbA1c≥7.0%, and FPG>7.0 mmol/L, but <13.9 mmol/L or 2hPG>11.1 mmol/L
* Informed consent has been signed
* Dampness and Heat in Spleen

Exclusion Criteria:

* The patients accepted diabetic treatment for more than a month continuously
* The patients were treated by drugs in 3 week before they were given test drugs
* Diabetic ketosis, diabetic ketoacidosis or serious inflammation in a month
* The contractive pressure >160 mmHg or diastolic pressure >100 mmHg
* Pregnant, preparing for pregnancy or breast-feeding women
* Mental patients
* The patients whose ALT or AST are >100U/L,and BUN or Cr are abnormal.
* The patients who have serious heart, lung, liver, kidney and brain or other primary complications
* Allergic persons
* The patients who are attending other clinical trial
* The patients who have serious diabetic complications
* The patients who ever attended this clinical trial
* Alcohol and / or psychoactive substances, drug abuse and dependency
* The person maybe loss for some reason such as work or life condition according to the investigator's judgement
* The lipid-lowering or antihypertensive drug dosage and category which the patients are taking could not be kept stable
* The patients who are eating some drugs or health food which can affect the body weight

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2010-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 12 weeks after treatment

SECONDARY OUTCOMES:
Fasting plasma glucose (FPG)、postprandial 2 hours plasma glucose(2hPG) | 12 weeks after treatment
blood and urine and stool routine examination, electrocardiogram (ECG)and liver and kidney function tests | 12 weeks after treatment
Ins(0h,1h,2h),blood lipids | 12 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Lin Tong, Ph.D, Study Chair — Guang' anmen Hospital of China Academy of Chinese Medical Sciences
Locations (4):
- China (4):
  - Beijing Traditional Chinese Medicine Hospital of the Capital University of Medical Sciences, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Ji Shui Tan Hospital of Beijing, Beijing, Beijing Municipality
  - Dongzhimen Hospital Attached to Beijing Traditional Chinese Medicine University, Beijing, Beijing Municipality